CLINICAL TRIAL: NCT01172704
Title: HIV/AIDS, Severe Mental Illness and Homelessness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Brady, Director, Mental Health Counseling & Behavioral Medicine Program Associate Professor of Psychiatry Boston University School of Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BMC HIV Prevention
Record Dates: First submitted 2010-06-09; First posted 2010-07-30 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: HIV; AIDS
Keywords: Motivational Interviewing; Serious Mental Illness; HIV/AIDS; HIV Testing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care as Usual (Active Comparator): Participants randomized to CAU receive the standard care given to patients of the Boston Medical Center who are interested in learning more about HIV/AIDS. Included in this care would be referrals for HIV counseling and testing.
  Interventions: Behavioral: Skills Building - Motivational Interviewing
- Skills Building - Motivational Interviewing (Experimental): Participants randomized to SB-MI will receive three individual sessions and a booster. Content of the sessions are as follows; Session 1: Risk Behavior Feedback & Building Motivation; Session 2: Building Motivation & Skill Selection and Practice; Session 3: Developing Change Plan & Skill Practice and Booster Session(s): Review Change Plan Implementation, Maintaining Motivation & Skill Practice.
  Interventions: Behavioral: Skills Building - Motivational Interviewing

INTERVENTIONS:
Behavioral: Skills Building - Motivational Interviewing — SB-MI incorporates Motivational Interviewing strategies into a psycho-educational HIV risk reduction protocol to help participants identify high-risk behaviors, reduce ambivalence about these behaviors, increase motivation to change behaviors, and develop a specific plan of action for risk reduction. Consistent with MI, information gathered at baseline regarding HIV risk behaviors is systematically reviewed in a personalized way with each participant at the outset of the intervention. This is designed to engage participants in becoming active agents in the change process and to assist participants in recognizing discrepancies between their current risk behaviors and goals and values, which typically do not include HIV infection or transmitting HIV to others. Also consistent with the principles of MI, participants are empowered to choose those educational and skills-based modules which "fit" their personal risk profile and values.

SUMMARY:
This is a two-arm randomized controlled trial (RCT) for 308 seriously mentally ill adults (SMI) engaging in risky sexual and/or drug use behavior, comparing a brief HIV primary and secondary prevention intervention [Skills building and Motivational Interviewing (SB-MI) to Care as Usual (CAU)]. The study setting is a large urban safety net Medical Center and outcomes will be measured at 3, 6, and 12 months. The SB-MI intervention (3 sessions + booster) was initially developed as the experimental condition in an R34 pilot project which demonstrated its feasibility and promise. For the proposed project, the investigators will recruit a larger sample which includes men and women with and without HIV, from various ethnic and racial groups, sexual orientations and housing arrangements, as well as a range of psychiatric disorders and functional capacities. In this way the investigators can more rigorously demonstrate the promise of SB-MI with SMI. The investigators will also conduct a sub-study after the 6 month follow-up to examine the impact at 12 months of an additional booster session for SB-MI participants. The investigators specific aims are:

1. To examine the effectiveness of a brief, tailored primary and secondary risk reduction strategy to CAU for people with serious mental illness. The desired outcomes include:

   * Decreased frequency of risk behaviors (number of partners, number of encounters)
   * Increased use of barrier precautions and IV needle cleaning
   * Positive changes in information and motivation, as well as risk behaviors
   * Increased HIV Counseling and Testing for those who do not know their HIV status
2. To examine the effectiveness of a 2nd booster session after the 6 month follow-up for ½ of participants randomized to SB-MI. The primary outcome will be:

   * Decreased frequency of risk behaviors and increased use of barrier precautions at the 12 month follow-up

DETAILED DESCRIPTION:
Our long-term objective is to reduce the incidence of HIV risk behavior for SMI by developing an intervention that can be easily translated and adapted to "real world" settings. Our proposed project is designed to augment previously-developed research on HIV risk reduction interventions for SMI. The innovations the investigators have developed include: 1) SB-MI intervention design that can be utilized with diverse participants with SM in contrast to other research which has focused on either primary or secondary prevention with a fairly discrete population, such as women of color, patients in a drug recovery program etc. The investigators will examine treatment response as a function of diverse participant characteristics; 2) SB-MI intervention is delivered in an individual format to provides a flexible structure for tailoring strategies and techniques for each participant's complex cognitive and psychosexual functioning, as well as his/her needs and values in contrast to research on HIV prevention in SMI which generally occurs in group and does not allow for individualized tailoring. In addition, our experience with group interventions is they do not easily allow for discussions of risk related to complex sexual and physical abuse histories, sex trading and other stigmatized activities characteristic of SMI. Our individualized approach affords maximum flexibility and privacy in selecting topics of intervention, which the investigators also believe to be essential to the spirit of Motivational Interviewing; 3) Previous interventions have typically been either very brief (e.g. one half-hour session) or time-intensive. In contrast, our intervention (3 sessions + 1 or 2 Booster(s)) is long enough to allow participants to form a working alliance with providers, but not so lengthy as to be burdensome or non-translatable for the real-world settings in which patients routinely seek care such as urban safety net Medical Center's; 4) a review of the literature suggests that many health behavior changes fade within a fairly short period of time; our inclusion of booster session and a sub-study examining the effect of a 2nd booster after the 6 month follow-up is a novel way of strengthening the effects of our intervention. The investigators will also be extending our follow-up period to 12 months, to allow us to further assess long-term change; and 5) No study to date has examined HIV counseling and testing as an outcome for this population (Senn & Carey, 2009). The investigators believe this represents a significant deficit in attending to the needs of SMI, given that testing and access to life-extending treatment should be an essential component to prevention interventions for SMI. Both our SB-MI and CAU conditions will include referrals for HIV testing where indicated, although the SB-MI intervention systematically supports motivation for participants seeking HIV counseling and testing services, whereas CAU provides information and general support for testing. The investigators hope to see that the attention paid to this issue in SB-MI yields greater access to HIV testing services.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for a serious mental illness (SMI)
* Engaged in HIV risk behavior during the previous 3 months
* Able to attend assessment and intervention appointments
* Have receptive and expressive English language skills sufficient for meaningful participation
* Are 19 years of age or older.
* Capable of providing informed consent.

Exclusion Criteria:

* Unable to comprehend the assessment and/or intervention materials.
* Unable to provide independent consent and/or under a full guardianship.
* Do not meet criteria for a serious mental illness (SMI)
* Have not engaged in HIV risk behavior during the previous 3 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-10; Primary Completion 2015-04 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Frequency of Risk Taking Behavior | One year
  Mean Changes from baseline to follow-ups at 6 and 12 months for constructs of the IMB (Information Motivation Behavior) Model will be larger for participants randomized to the SB-MI condition compared to CAU.

SECONDARY OUTCOMES:
HIV Counseling & Testing | One year
  Participants in SB-MI will demonstrate higher rates of accessing HIV counseling and testing at 6 month follow-up, as compared to participants in CAU.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Brady, PhD, Principal Investigator — Boston University; Jori Berger-Greenstein, PhD, Study Director — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States